CLINICAL TRIAL: NCT03349957
Title: Retrospective Study on TACE for HCC by TANDEM and Idarubicin
Brief Title: TACE for HCC by TANDEM and Idarubicin
Acronym: TANDEM-IDA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0390
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2017-11

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Idarubicin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Transarterial chemoembolization using TANDEM and idarubicin — Transarterial chemoembolization using TANDEM and idarubicin

SUMMARY:
DcBeads and lipiodol-transarterial chemoembolization (TACE) of hepatocellular carcinoma (HCC) using doxorubicin result in about 50% objective response rate at 6 months (Precision V study, Lammer et al. CVIR 2010) We previously demonstrated that idarubicin was the most effective drug on 3 HCC cell lines (Boulin et al., Anticancer drugs 2009). We tested idarubicin-loaded beads in a phase I trial (Boulin et al., Aliment Pharmacol Therapy 2012) and more recently in a prospective multicentric phase II trial (IDASPHERE II, Magna Cum Laude CIRSE 2017, B Guiu et al.). This trial was stopped at interim analysis because the endpoint was reached.

Tandem beads are precisely calibrated, of small size, allowing the maximization of ischemic effects together with an optimal efficacy of the drug. We previously published that idarubicin was able to load fastly in Tandem, with minimal modification of bead diameter and a very interesting releasing profile of the drug (Guiu et al., JVIR 2015).

We used TANDEM combined with idarubicin in our practice for the treatment of HCC by TACE (in-label use of beads and the drug).

No clinical study (even retrospective) has been published so far with TANDEM-IDA (except our first paper published in JVIR in 2015, only 4 patients).

Here we propose to collect the retrospective data of patients treated by TANDEM-IDA, to help to design a future multicentric randomized phase II trial

ELIGIBILITY:
Inclusion Criteria:

HCC according to histological examination or Barcelona criteria Measurable targets according to mRECIST v1.1 Child A or B7 cirrhosis (without decompensation in the past 6 months) HCC not candidate to surgery or ablation Age ≥ 18 years Performance status 0 or 1 Thrombocytes ≥ 50 000/mm3, neutrophil count≥ 1 000/mm3, creatininemia ≤ 150 µmol/L No cardiac failure

Exclusion Criteria:

Follow-up < 1month Lobar/main portal venous thrombus Prior treatment by systemic chemotherapy or radioembolization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by TACE for HCC by TANDEM and idarubicin
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
tumeur response | 1 day
  tumeur response

CONTACTS AND LOCATIONS:
Overall Officials: Boris GUIU, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC